CLINICAL TRIAL: NCT07304544
Title: Study on the Impact of Roy Adaptation Model Nursing on Psychological State and Quality of Life of Post-Colostomy Patients and Exploration of Its Mechanism
Brief Title: Roy Adaptation Model in Post-Colostomy Care: Mind & Life Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WestChinaH-SJ-2025-01
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Colostomy Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): On the basis of routine nursing, RAM-based nursing was implemented for 12 weeks
  Interventions: Behavioral: RAM-based nursing
- Control group (No Intervention): Received routine post-colostomy nursing for 12 weeks: (1) Stoma care: Guidance on stoma cleaning, ostomy bag replacement, and observation of stoma color and secretion; (2) Physiological care: Pain management, dietary guidance, and prevention of postoperative complications (e.g., infection, constipation); (3) Routine health education: Distribution of stoma care manuals and brief psychological comfort.

INTERVENTIONS:
Behavioral: RAM-based nursing — On the basis of routine nursing, RAM-based nursing was implemented for 12 weeks
  Arms: Intervention Group

SUMMARY:
The goal of this randomized controlled trial is to learn if the Roy Adaptation Model (RAM) nursing program improves anxiety, depression, and quality of life in adults who have recently received a colostomy. It will also learn about changes in stress and inflammation-related blood markers. The main questions it aims to answer are:

Does 12-week RAM nursing lower anxiety and depression scores compared with routine nursing? Does RAM nursing raise quality-of-life scores and beneficially alter blood levels of cortisol, IL-6, TNF-α, serotonin, and dopamine? Researchers will compare RAM nursing (one-to-one education, cognitive-behavioral support, family training, and phone follow-up) to routine stoma-care education only.

Participants will:

Receive either RAM nursing or routine nursing for 12 weeks Complete anxiety, depression, and quality-of-life questionnaires at baseline and week 12 Provide blood samples at baseline and week 12 to measure stress and inflammation markers (which was a routine test for normal colostomy patients)

ELIGIBILITY:
Inclusion Criteria:

* Underwent elective colostomy (permanent or temporary) due to colorectal cancer, inflammatory bowel disease, or intestinal obstruction;
* Postoperative time ≤ 1 week;
* Age 18-75 years;
* Consciousness clear, able to communicate normally and complete questionnaire surveys;
* Voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

* Complicated with severe cardiovascular, liver, kidney, or mental diseases;
* History of anxiety, depression, or other mental disorders before surgery;
* Stoma complications (e.g., stoma prolapse, ischemia, infection) requiring reoperation;
* Loss to follow-up or refusal to cooperate with the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Self-Rating Anxiety Scale (SAS) score | Week 12
  Sum the scores of all 20 items. The total score ranges from 20 to 80. A cut-off score of 50 indicates significant anxiety,the higher the score,the higher the anxiety level (scores ≥50 suggest anxiety symptoms).
Self-Rating Depression Scale (SDS) | 12 weeks
  Sum the scores of all 20 items. The total score ranges from 20 to 80. A cut-off score of 53 indicates significant depression. The higher the score, the depression level is higher(scores ≥53 suggest depressive symptoms).

SECONDARY OUTCOMES:
World Health Organization Quality of Life-Brief Interpretation(WHOQOL-BREF) scores | Week 12
  1. Reverse Scoring: For item 6 (pain/discomfort), reverse the score (1=5, 2=4, 3=3, 4=2, 5=1) because higher scores on this item indicate poorer quality of life. All other items are scored as per the original response.
  2. Domain Scores: Calculate the average score for each domain (Physical Health: Items 1-8; Psychological Health: Items 9-14; Social Relationships: Items 15-17; Environmental Domain: Items 18-26).
  3. Standardization: Convert each domain average score to a standard score (0-100) using the formula: Standard Score = [(Average Score - 1) / 4] × 100. Higher standard scores indicate better quality of life in that domain.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No